CLINICAL TRIAL: NCT07304986
Title: A Novel Method for Evaluating i-PRF Usage in Vestibular Socket Therapy for Immediate Implant in Defective Fresh Extraction Site
Brief Title: Efficacy of i-PRF Usage in Vestibular Socket Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdallah Mohmmed Elshamy, Assistant lecturer of periodontology, Al-Azhar University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 921/1704
Record Dates: First submitted 2024-07-31; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Esthetic Zone
MeSH Terms: interventions — proliferation regulatory factors, human urine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- deficient facial plate of bone management VST only (Experimental): Sockets with deficient facial plate of bone and intact soft tissue will receive VST only.
  Interventions: Procedure: Immediate implant with VST
- deficient facial plate of bone management with VST and iPRF. (Active Comparator): Sockets with deficient facial plate of bone and intact soft tissue will receive VST and iPRF.
  Interventions: Procedure: Immediate implant with VST and i-prf

INTERVENTIONS:
Procedure: Immediate implant with VST — Preoperative procedure: cone beam computed tomography (CBCT) scan will be used for diagnosis and treatment planning. Nonsurgical periodontal treatment including scaling and root planning will be performed as needed. Under local anesthesia sulcular incisions will be made, and then hopeless teeth will be extracted atraumatically using periotomes. Socket lavage and curettage will be done thoroughly, and dental implants will be inserted.
  Arms: deficient facial plate of bone management VST only
Procedure: Immediate implant with VST and i-prf — Preoperative procedure: cone beam computed tomography (CBCT) scan will be used for diagnosis and treatment planning. Nonsurgical periodontal treatment including scaling and root planning will be performed as needed. Under local anesthesia sulcular incisions will be made, and then hopeless teeth will be extracted atraumatically using periotomes. Socket lavage and curettage will be done thoroughly, and dental implants will be inserted with i-prf.
  Arms: deficient facial plate of bone management with VST and iPRF.

SUMMARY:
This study aims for evaluation of A novel method for evaluating i-PRF usage in vestibular socket therapy for immediate implant in defective fresh extraction site.

DETAILED DESCRIPTION:
The ultimate objective of implant treatment is providing long-lasting, healthy hard and soft tissue architecture while minimizing intraoperative surgical trauma and postoperative complications. Reducing treatment duration and providing a predictable esthetic outcome are fundamental. Immediate implant placement in fresh extraction sockets is an appealing treatment option satisfying many of these requirements. However, a major concern with immediate implant placement is the possible resorption of the facial bone plate as indicated in multiple studies. This, in turn, results in loss of proper soft tissue support, thus compromising the final esthetic outcome of the implant- supported restoration. Furthermore, post extraction bone resorption would be compounded by the presence of a thin or preexisting facial bone defect and/or a thin gingival phenotype. Multiple approaches were suggested to prevent facial bone resorption and optimize the final esthetic outcome after immediate implant placement in sockets with intact facial bone and soft tissue. These approaches include simple ones like applying a graft in the gap between the implant and the facial socket wall and more sophisticated approaches such as the socket shield technique . The presence of bone and/or soft tissue defects after tooth extraction is not an uncommon finding, further complicating immediate implant placement. Several classifications for fresh extraction sockets were proposed to facilitate the selection of optimum treatment for individual cases.

Currently, a serious of studies has shown that iPRF can produce significantly greater concentrations of platelets and leukocytes when compared to the L-PRF and A-PRF.

ELIGIBILITY:
Inclusion Criteria:

* Patients has one hopeless tooth in the maxillary anterior region with TYPE II according to Elian classification of sockets (10) and sufficient bone apically and palatally.
* The presence of a natural contralateral tooth for the tooth being replaced.

Exclusion Criteria:

* Extraction sockets were grade III.
* Acute infection related to hopeless tooth.
* Allergy to any material or medication used in the study.
* Medically compromised patients according to modified Cornell Medical Index.
* Heavy smokers.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2026-01-21 (Estimated); Study Completion 2026-03-21 (Estimated)

PRIMARY OUTCOMES:
assessment of pink aesthetic score of the gingiva | 6 and 9 months.
  Assessment of clinical and aesthetic parameters after the newly proposed immediate implant placement technique. using pik aesthetic score of gingiva, The Pink Esthetic Score (PES) is a dental assessment tool scoring gingival aesthetics around implants, evaluating mesial/distal papillae, tissue level/contour/color/texture, and alveolar deficiency.
  Scoring System 0 (Poor): Marked deficiency or abnormality.
  1. (Fair): Slight change or minor discrepancy.
  2. (Excellent): Healthy, normal, ideal appearance.

SECONDARY OUTCOMES:
Facial bone thickness | base line, 6 and 9 months.
  Assessment of radiographic parameters after the newly proposed immediate implant placement technique.will be assessed from implant surface to outer surface of bone will be recorded using cone beam CT, at base line, 6 and 9 months. and will be recorded in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: abdullah el-shamy, MSC, Principal Investigator — Al-Azhar University
Locations (1):
- AlAzharU, Cairo, Nasr City, Egypt